CLINICAL TRIAL: NCT00749528
Title: Sectional Prospective Randomised Study of Evaluation Toxic Metals, Trace Elements Status and Total Antioxidant Activity in Children With Recurrent Wheezing.
Brief Title: Evaluation of Toxic Metals, Trace Elements and Total Antioxidant Activity in Children With Recurrent Wheezing
Status: Completed | Type: Observational
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Cem Hasan Razi, Kecioren Education and Training Hospital, Kecioren Education and Training Hospital
Other Study IDs: 2008-08-11
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2008-08

CONDITIONS: Asthma; Wheezing
Keywords: Wheezing; Hair trace elements; Hair toxic metals; Oxidative stress
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Group 1: Children with recurrent wheezing. Plasma and Hair specimen are retined Group 2: Healthy children. Plasma and Hair specimen are retined
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Children vith recurrent wheezing
- 2: Healthy children

SUMMARY:
The purpose of this study is to evaluate hair trace elements and toxic metals and plasma total antioxidant activity in children with recurrent wheezing and to evaluate whether these toxic metals and trace elements have any impact on serum cytokine levels.

DETAILED DESCRIPTION:
Context:

In many studies it was demonstrated that children are much more susceptible than adults for environmental toxic metal exposure. Hair analysis is a promising tool for routine clinical screening and diagnosis of heavy metal exposure and essential trace element states in the human body. Additionally it was demonstrated that oxidants and antioxidants play a central role in the pathogenesis of many pulmonary diseases including asthma. Furthermore, toxic metals, trace elements and oxidative stress have many pivotal role on immune system.

Objective:

To evaluate and compare hair toxic metals, hair essential trace elements levels and plasma total antioxidant activity between children with recurrent wheezing and age and sex matched healthy children.

Intervention: Hair samples will be collected for the analysis of the toxic metals, trace elements. Blood samples will be collected for the analysis of the cytokine levels and plasma antioxidant activity.

Study Measures:

Differences in hair toxic metals, hair trace elements, plasma cytokine levels and plasma total antioxidant activity will be compared between children with recurrent wheezing and age-sex matched healthy children

ELIGIBILITY:
Inclusion Criteria:

* Children with recurrent wheezing ages between 6 months to 6 years old.
* Age and sex matched healthy children for control group.
* Parental/guardian permission (informed consent)

Exclusion Criteria:

* Systemic corticosteroid use in the last 30 days
* Chronic lung diseases including cystic fibrosis
* Immunodeficiency
* Known renal or hepatic dysfunction
* Respiratory truck infections in the last 30 days
* Anatomic abnormalities of the respiratory tract
* Suspected foreign body aspiration or croup
* Immunosuppressive or immunostimulant treatment

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Group 1: Children with recurrent wheezing Group 2: Age and sex matched healthy children
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Hair toxic metal and trace element status in the two groups | 6 months

SECONDARY OUTCOMES:
To compare plasma total antioxidant activity in the two groups. | 6 months
Effect of heavy metals and trace elements on plasma cytokine levels and difference between the two groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: C H RAZI, MD, Study Director — Kecioren Education and Training Hospital; C H RAZI, MD, Principal Investigator — Kecioren Education and Training Hospital
Locations (1):
- Kecioren Eğitim Araştırma Hastanesi, Ankara, Kecioren, Turkey (Türkiye)